CLINICAL TRIAL: NCT03358212
Title: Safety and Efficacy of Post-operative Denosumab Strategy for Giant Cell Tumor of Bone Treatment in China：Correlation Between Recurrence and Drug Withdrawl
Brief Title: Safety and Efficacy of Post-operative Denosumab Strategy for Giant Cell Tumor of Bone Treatment in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, GUO WEI, Chief of Musculoskeltal Tumor Center, Peking University People's Hospital
Other Study IDs: GCTB-China
Record Dates: First submitted 2017-11-26; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Giant Cell Tumor of Bone
Keywords: giant cell tumor of bone; Denosumab; post-operative
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Denosumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- denosumab used postoperatively: the postoperative denosumab group, including patients receiving denosumab after piecemeal intralesional curettage aided by digital subtraction angiography(DSA) and balloon occlusion of abdominal aorta;
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — Denosumab 120mg was administrated to patients by subcutaneous injection every four weeks, with loading doses on Day 8 and Day 15 of the first cycle.Patients were instructed to take calcium supplements orally every day and avoid any oral operation during treatment
  Other Names: XGEVA

SUMMARY:
This prospective observational study is going to figure out the safety and efficacy of denosumab as an post-operative strategy.All the patients enrolled will take denosumab according to the protocols.We focus on the recurrence rate after the drug withdrawl and possibility of malignant transformation.

DETAILED DESCRIPTION:
This prospective observational study is going to figure out the safety and efficacy of denosumab as an post-operative strategy.

This study only included patients who meet all the following criteria: (1) With treatment-naïve sacral giant-cell tumor (GCT) firstly treated in our center (for referral patients, only those with definite diagnosis were included); (2) Being diagnosed with classic giant-cell tumor of bone (GCTB) by puncture pathology prior to treatment (for referral patients, definite diagnosis shall be made by the Pathology Department in our center through pathology consultation on tissue sections); (3) previously denosumab-naïve.

Data collection:The following data of patients included in this study were collected: (1) basic information: age, gender; (2) pathological data: puncture pathological diagnosis, and postoperative pathological findings; (3) the imaging findings (including X-ray, CT, Magnetic resonance(MR), Positron Emission Tomography-Computed Tomography(PET-CT)) and functional assessment of patients in the neoadjuvant denosumab group before and after the use of denosumab; (4) intraoperative blood loss, and duration of operation; (5) imaging findings in postoperative follow-up re-examination and outcome.

functional assessment: For sacral giant cell tumor:The Motor Urination defecation(MUD) scoring system published on Spine by our center in 2016 , which include three domains (motor function and sensation of lower limbs [M], urination and uriesthesia [U], and Defecation and rectal sensation [D]) with three items in each domain (each item can be scored by 0, 1, 2 or 3, and the maximum score is 27), was applied in the functional assessment of sacral nerves.

For GCT occurs in Limbs ,we use Musculoskeletal Tumor Society (MSTS) 93 to record the function.

All the patients enrolled will take denosumab according to the protocols:denosumab 120mg was administrated to patients by subcutaneous injection every four weeks, with loading doses on Day 8 and Day 15 of the first cycle,them take it monthly till 1 year after the surgery.We focus on the recurrence rate after the drug withdrawl and possibility of malignant transformation.

ELIGIBILITY:
Inclusion Criteria:

(1) With treatment-naïve sacral GCT firstly treated in our center (for referral patients, only those with definite diagnosis were included); (2)single center lesion (3) Being diagnosed with classic GCTB by puncture pathology prior to treatment (for referral patients, definite diagnosis shall be made by the Pathology Department in our center through pathology consultation on tissue sections); (4) previously denosumab-naïve.

Exclusion Criteria:(1)primary malignant giant cell tumor of bone(2)radiation therapy in history(3)lung metastasis at first diagnosis

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with giant cell tumor of bone referred to, or being treated at Peking University People's Hostpital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
recurrence without metastasis | up to 2 years
  CT or MR proof that the tumor relapse in the primary site by at least two radiologist

SECONDARY OUTCOMES:
metastasis without recurrence | up to 2 years
  confirmed via lung CT scan by at least two radiologist
death from other disease | up to 2 years
  patient die from another disease but must not from giant cell tumor
death from giant cell tumor | up to 2 years
  patient die from the tumor itself

CONTACTS AND LOCATIONS:
Overall Officials: Guo Wei, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutkowski P, Ferrari S, Grimer RJ, Stalley PD, Dijkstra SP, Pienkowski A, Vaz G, Wunder JS, Seeger LL, Feng A, Roberts ZJ, Bach BA. Surgical downstaging in an open-label phase II trial of denosumab in patients with giant cell tumor of bone. Ann Surg Oncol. 2015 Sep;22(9):2860-8. doi: 10.1245/s10434-015-4634-9. Epub 2015 Jun 2. PMID 26033180
- [Background] Mak IW, Evaniew N, Popovic S, Tozer R, Ghert M. A Translational Study of the Neoplastic Cells of Giant Cell Tumor of Bone Following Neoadjuvant Denosumab. J Bone Joint Surg Am. 2014 Aug 6;96(15):e127. doi: 10.2106/JBJS.M.01332. PMID 25100780
- [Background] Ueda T, Morioka H, Nishida Y, Kakunaga S, Tsuchiya H, Matsumoto Y, Asami Y, Inoue T, Yoneda T. Objective tumor response to denosumab in patients with giant cell tumor of bone: a multicenter phase II trial. Ann Oncol. 2015 Oct;26(10):2149-54. doi: 10.1093/annonc/mdv307. Epub 2015 Jul 23. PMID 26205395
- [Background] Branstetter DG, Nelson SD, Manivel JC, Blay JY, Chawla S, Thomas DM, Jun S, Jacobs I. Denosumab induces tumor reduction and bone formation in patients with giant-cell tumor of bone. Clin Cancer Res. 2012 Aug 15;18(16):4415-24. doi: 10.1158/1078-0432.CCR-12-0578. Epub 2012 Jun 18. PMID 22711702
- [Background] Wojcik J, Rosenberg AE, Bredella MA, Choy E, Hornicek FJ, Nielsen GP, Deshpande V. Denosumab-treated Giant Cell Tumor of Bone Exhibits Morphologic Overlap With Malignant Giant Cell Tumor of Bone. Am J Surg Pathol. 2016 Jan;40(1):72-80. doi: 10.1097/PAS.0000000000000506. PMID 26414220
- [Background] Chawla S, Henshaw R, Seeger L, Choy E, Blay JY, Ferrari S, Kroep J, Grimer R, Reichardt P, Rutkowski P, Schuetze S, Skubitz K, Staddon A, Thomas D, Qian Y, Jacobs I. Safety and efficacy of denosumab for adults and skeletally mature adolescents with giant cell tumour of bone: interim analysis of an open-label, parallel-group, phase 2 study. Lancet Oncol. 2013 Aug;14(9):901-8. doi: 10.1016/S1470-2045(13)70277-8. Epub 2013 Jul 16. PMID 23867211